CLINICAL TRIAL: NCT03137212
Title: Study of Safety and Efficacy of Percutaneous Coronary Intervention Combined With Thrombolysis by Recombinant Human Prourokinase at Different Time
Brief Title: Safety and Efficacy of Percutaneous Coronary Intervention Combined With Thrombolysis at Different Time
Acronym: SEPCIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SecondJilinU-2
Record Dates: First submitted 2017-04-16; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Acute ST Segment Elevation Myocardial Infarction
Keywords: Percutaneous Coronary Intervention; STEMI; Thrombosis
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Thrombosis | interventions — Fibrinolytic Agents

STUDY DESIGN:
Intervention Model Description: The patients with STEMI will be divided into two group randomly. Patients of A group will be treated by thrombolysis and then 3-6 hours will be treated by PCI. Patients of B group will be treated by thrombolysis and then 6-24 hours will be treated by PCI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A group (Experimental): STEMI patients first are given thrombolysis and then transfer to PCI center to be treated by PCI 3-6 hours after thrombolysis if the thrombolysis is successful. if the thrombolysis is not successful, patients will be treated by PCI immediately.
  Interventions: Combination Product: thrombolysis and PCI of A type
- B group (Experimental): STEMI patients first are given thrombolysis and then transfer to PCI center to be treated by PCI 6-24 hours after thrombolysis if the thrombolysis is successful. if the thrombolysis is not successful, patients will be treated by PCI immediately.
  Interventions: Combination Product: thrombolysis and PCI of B type

INTERVENTIONS:
Combination Product: thrombolysis and PCI of A type — STEMI patients first are given thrombolysis and then transfer to PCI centers to be treated by PCI 3-6 hours after thrombolysis.
  Arms: A group
Combination Product: thrombolysis and PCI of B type — STEMI patients first are given thrombolysis and then transfer to PCI centers to be treated by PCI 6-24 hours after thrombolysis.
  Arms: B group

SUMMARY:
Patients with acute ST-segment elevation myocardial infarction and thrombolysis indications, will be given the recombinant human prourokinase for thrombolysis treatment, and in accordance with the guidelines, will be treated with coronary angiography examination 3 to 24 hours after thrombolysis. The study will explore the best time for interventional therapy combined with thrombolysis.

DETAILED DESCRIPTION:
The noninferiority multicenter, prospective, randomized, controlled study of urokinase of restructuring the original design evaluation (rhPro - UK) at different times after thrombolysis combined with percutaneous coronary intervention（PCI）therapy of acute ST segment elevation myocardial infarction.Patients with acute ST segment elevation myocardial infarction and thrombolysis indications, will be given the recombinant human prourokinase for thrombolysis treatment, and in accordance with the guidelines, will be treated with coronary angiography examination 3 to 24 hours after thrombolysis. The study will explore the best time for interventional therapy combined with thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 to 70 years old, gender not limited
* 30 minutes or more persistent ischemia chest pain, and symptoms can't ease by treated by nitroglycerin
* In two or more lead ecg ST-segment（the line between QRS complex finish point and the start point of T wave in electrocardiogram) elevation ≥ 0.1mv, or two or more than two neighboring chest lead ST-elevation ≥0.2mv
* Persistent ischemia chest pain less than 6 hours, door to balloon time>90 minutes and transfer time >120 minutes
* Accept coronary arteriography and intervention treatment
* Signed informed consent

Exclusion Criteria:

* Pregnancy and lactation, menstrual period women
* Blood disease, clotting hemorrhagic disease, any part of active bleeding or bleeding tendency physique
* History of trauma in two months, including biopsy and received surgical operation
* History of the great vessels punctured in two weeks that could not oppression
* History of ischemic or hemorrhagic stroke and cerebrovascular accident
* Cardiac shock,reinfarction again, right ventricular myocardial infarction, history of cardiopulmonary resuscitation (CPR)
* History of PCI or coronary artery bypass grafting（CABG）
* Killip classification level III（a standard of heart function classification） or above, or cardiac mechanical complications such as cardiac rupture
* History of eyeground hemorrhage
* Currently use of therapeutic doses of anticoagulants, such as warfarin, etc
* Uncontrolled hypertension, systolic blood pressure before thrombolysis is still 160 mmHg or higher, diastolic blood pressure is still 100 mmHg or higher
* Active internal bleeding (such as gastrointestinal bleeding), urogenital system, or have not cure of peptic ulcer in four weeks
* Severe liver and kidney dysfunction
* Intracranial tumor, suspicious aortic dissection, arteriovenous malformation, aneurysm
* Thrombolysis treatment in one week
* Allergies of thrombolysis drug or contrast
* Participated in any clinical trials within three months

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-04-17 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Post-PCI（percutaneous coronary intervention） myocardial perfusion (TIMI flow grade) | intraoperative
  The investigators will check myocardial perfusion (TIMI flow grade) after PCI （percutaneous coronary intervention）immediately.
The incidence of no reflow | intraoperative
  The investigators will check the incidence of no reflow after PCI（percutaneous coronary intervention） immediately.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events （MACE） | 1 month, 3 month,6 month,12 month
  Death and recurrence of myocardial infarction and target vessels revascularization
Post-PCI heart function | 1 month, 3 month,6 month,12 month
  The value of ejection fraction will be examined by cardiac ultrasound for heart function.
The incidence of serious bleeding events | 1 year
  The incidence of serious bleeding events including all cause.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Liu, Doctor, Principal Investigator — Second Hospital of Jilin University
Locations (1):
- The second hospital of Jilin university, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
when the investigators complete the study and publish our data